CLINICAL TRIAL: NCT03717987
Title: The Effect of Botulinum Toxin A In Patients With Excessive Gingival Display With And Without Zinc Supplementation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Mohamed Fouad Shemais, Demonstrator at Faculty of Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 130388
Record Dates: First submitted 2018-10-21; First posted 2018-10-24 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Excessive Gingival Display
Keywords: gummy smile; Botulinum toxin type A; excessive gingival display
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulinum toxin A injection (Active Comparator): Botulinum toxin type A will be injected in all patients at both sides into the "Yonsei point," (3Units) the point that would target 3 muscles responsible for upper lip elevation during smiling, including the LLSAN, in a single injection. This landmark was identified as the center of a triangle formed by the convergence of the LLSAN, the LLS, and the Zminor muscles and is located 1 cm lateral to the ala horizontally and 3 cm above the lip line vertically in both men and women.
  Interventions: Drug: Botulinum toxin type A
- Zinc supplementationj prior to Botulinum toxin A injection (Active Comparator): Patients in the intervention group will take zinc supplement tablets to increase zinc levels for 4 days before botulinum toxin injections. While patients in the control group will take placebo tablets 4 days prior to the injections. All tablets will be placed in envelopes for blinding the operator, and numbered by a supervisor to allocate patients again in their groups for statistical results. Botulinum toxin type A will be injected in all patients at both sides into the "Yonsei point," (3Units) the point that would target 3 muscles responsible for upper lip elevation during smiling, including the LLSAN, in a single injection. This landmark was identified as the center of a triangle formed by the convergence of the LLSAN, the LLS, and the Zminor muscles and is located 1 cm lateral to the ala horizontally and 3 cm above the lip line vertically in both men and women.
  Interventions: Drug: Botulinum toxin type A; Dietary Supplement: Zinc supplementation

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum toxin type A will be injected in all patients at both sides into the "Yonsei point," (3Units) the point that would target 3 muscles responsible for upper lip elevation during smiling, including the LLSAN, in a single injection. This landmark was identified as the center of a triangle formed by the convergence of the LLSAN, the LLS, and the Zminor muscles and is located 1 cm lateral to the ala horizontally and 3 cm above the lip line vertically in both men and women (Hwang et al. 2009) and (Nasr et al. 2015).
Dietary Supplement: Zinc supplementation — zinc supplementation will be given to patients in the intervention arm 4 days prior to Botulinum toxin type A injection
  Arms: Zinc supplementationj prior to Botulinum toxin A injection

SUMMARY:
It has been noted since the start of using botulinum toxin for both medical and cosmetic indications that some patients simply don't achieve the responses to the drug that others do, leading to increased dose requirements and more frequent treatments. It was from this observation that researchers started to look at the zinc levels of patients and consider the concept of supplementation. In a recent systematic review, it was reported that there is very scant evidence to determine the exact clinical effects and duration of BTX-A when injected to treat gummy smile patients. Therefore, the investigators want to administrate of zinc supplements to patients prior to BTX-A injection to study if it will enhance its clinical effects, since it is from the zinc dependent metalloprotease family, where for each botulinum toxin molecule to be effective in paralyzing a muscle response it must be associated with a molecule of zinc which could be found within the cells of the body.

Participants with esthetic concern of excessive gingival display who meets the inclusion criteria will be assigned randomly and blindly to one of the 2 groups. Patients in the intervention group will take zinc supplement tablets to increase zinc levels for 4 days before botulinum toxin injections. While patients in the control group will take placebo tablets 4 days prior to the injections. All tablets will be placed in envelopes for blinding the operator, and numbered by a supervisor to allocate patients again in their groups for statistical results. Botulinum toxin type A will be injected in all patients at both sides into the "Yonsei point," (3Units) the point that would target 3 muscles responsible for upper lip elevation during smiling, including the LLSAN, in a single injection. This landmark was identified as the center of a triangle formed by the convergence of the LLSAN, the LLS, and the Zminor muscles and is located 1 cm lateral to the ala horizontally and 3 cm above the lip line vertically in both men and women. After 2 weeks the patients would come for an additional touch up dose (1 unit at each injection point).

ELIGIBILITY:
Inclusion Criteria:

* Patients with excessive gingival display >3mm.
* Adults >18 years.
* Non-smokers.
* Systemically healthy.
* Normal clinical crown dimensions.
* Hypermobile lip and Short or mild VME.

Exclusion Criteria:

* Severe VME.
* Pregnant or lactating females.
* Patients with inflamed gingiva or gingival enlargement.
* Inflammation or infection at the site of injection.
* Patients with known allergy to any of the components of BTX-A or BTX-B (i.e. BTX, human albumin, saline, lactose and sodium succinate).
* Patients using anticholinesterase or other agents interfering with neuromuscular transmission.
* Psychologically unstable or who have questionable motives and unrealistic expectations.
* Dependent on intact facial movements and expressions for their livelihood (e.g. actors, singers, musicians and other media personalities).
* Afflicted with a neuromuscular disorder (e.g. myasthenia gravis, Eaton-Lambert syndrome).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Change in the amount of gingival display | it will be measured after 2 weeks, then after 6, 12, 18 and 24 weeks
  Change in gingival display will be measured using a ruler

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shemais N, Elarab AE, ElNahass H. The effect of botulinum toxin A in patients with excessive gingival display with and without zinc supplementation: randomized clinical trial. Clin Oral Investig. 2021 Nov;25(11):6403-6417. doi: 10.1007/s00784-021-03944-2. Epub 2021 May 5. PMID 33950373